CLINICAL TRIAL: NCT06006767
Title: Links Between Rhythmic Handwriting Deficits and General Rhythmic Abilities in Children With Developmental Coordination Disorder: a Pilot Study. TDC-Rythme
Brief Title: Rhythmic Handwriting Deficits and General Rhythmic Abilities in Children
Acronym: TDC-Rythme
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL23_0112
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Developmental Coordination Disorder
Keywords: : Developmental Coordination Disorder; Rhythm; Rhythmic skills; Handwriting
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with Developmental Coordination Disorder (DCD), a neurodevelopmental disorder that affects motor skills and motor learning (APA, 2013), have been reported to manifest rhythmic deficits in handwriting domain, as well as general rhythmic deficits (i.e., regardless handwriting context per se) (Rosenblum & Regev, 2013). Accordingly, children with DCD struggle in tasks like synchronising to an external musical rhythm (in rhythm production tasks) or even in discrimination tasks such as detecting beat deviations, i.e., in rhythm perception tasks (INSERM collective expertise, 2019).

These rhythmic deficits which manifest in a variety of tasks and conditions support the hypothesis of a "generalised dysrhythmia" in DCD, according to which the rhythmic deficits - in perceptual tasks and motor production - could have a common source, namely a mechanism devoted to rhythm processing (a cerebral mechanism involved in the perception of rhythm) and independent of the effectors involved and the type of task considered.

However, the nature of the relationships between general rhythmic skills (perceptual and motor) and rhythmic abilities when engaged in handwriting movement is largely unknown in DCD. Whether a common source drives these diverse rhythmic deficits remains to explore. If this hypothesis were to be confirmed, this would pave the way for innovative therapeutic tools (e.g., serious games) for training a central rhythmic processing mechanism (rhythm perception), which could positively impact in turn rhythmicity of thandwriting movement in this population.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7 to 10 inclusive
* Children who can read and write
* Diagnosis of DCD according to DSM-5 criteria (APA, 2015)
* Native French speaker
* Living with at least one parent

Exclusion Criteria:

* Intellectual development disorder confirmed or suspected during the initial evaluation phase in the MPEA department.
* Presence or suspected presence of a visual impairment at the root of the motor skills deficit.
* Presence or suspected presence of a neurological motor disorder (e.g. sensory impairment, cerebral palsy, muscular dystrophy, degenerative disease).
* Not affiliated to a social security scheme or not benefiting from such a scheme.
* Absence of written, informed consent from parents.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: DCD children
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2023-10-16 (Estimated); Primary Completion 2025-07-16 (Estimated); Study Completion 2026-01-17 (Estimated)

PRIMARY OUTCOMES:
The rhythm of handwriting movement | 1 day at First visit
  measured by the variability of the handwriting movement frequency, obtained by calculating the inverse of the period of the strokes (local minima of speed) from the children's writing productions on a graphic tablet (Danna et al., 2013).

SECONDARY OUTCOMES:
The rhythmic variables | 1 day at First visit
  Perceptual and motor rhythmic skills out of context of handwriting, obtained from the assessment of rhythmic skills using the gold-standard BAASTA battery (Dalla Bella et al., 2017).
Speed of handwriting : abnormal peak velocity fluctuations during handwriting movement | 1 day at First visit
  Abnormal variations of the speed peaks during the writing movement are processed from the raw or transformed data according to the same conditions as in BHK test condition depending on the normality or non-normality of data.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital La Colombière - CHU de Montpellier, Montpellier, France

REFERENCES:
- [Background] American Psychiatric Association (APA) (2013). Diagnostic and statistical manual of mental disorders (5th ed.). Arlington, VA: American Psychiatric Publishing.
- [Background] Dalla Bella S, Farrugia N, Benoit CE, Begel V, Verga L, Harding E, Kotz SA. BAASTA: Battery for the Assessment of Auditory Sensorimotor and Timing Abilities. Behav Res Methods. 2017 Jun;49(3):1128-1145. doi: 10.3758/s13428-016-0773-6. PMID 27443353
- [Background] Danna J, Paz-Villagran V, Velay JL. Signal-to-noise velocity peaks difference: a new method for evaluating the handwriting movement fluency in children with dysgraphia. Res Dev Disabil. 2013 Dec;34(12):4375-84. doi: 10.1016/j.ridd.2013.09.012. Epub 2013 Oct 18. PMID 24139714
- [Background] Expertise Collective INSERM (2019). Trouble développemental de la coordination ou dyspraxie, Paris : Les Editions EDP Sciences.
- [Background] Rosenblum S, Regev N. Timing abilities among children with developmental coordination disorders (DCD) in comparison to children with typical development. Res Dev Disabil. 2013 Jan;34(1):218-27. doi: 10.1016/j.ridd.2012.07.011. Epub 2012 Sep 6. PMID 22960066